CLINICAL TRIAL: NCT02891707
Title: Mobile Device Outcomes-based Rehabilitation Program
Acronym: MDORP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Walter Reed National Military Medical Center (U.S. Federal Agency); Uniformed Services University of the Health Sciences (U.S. Federal Agency); University of Miami (Other); Miami VA Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 407406
Record Dates: First submitted 2016-08-24; First posted 2016-09-07 (Estimated); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Transfemoral Amputation; Transtibial Amputation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Active Comparator): The investigators will recruit 20 healthy subjects at Walter Reed National Military Medical Center (WRNMMC) with the goal of consenting and enrolling 15 healthy subjects to assess the reliability and validity the wearable Rehabilitative Lower-limb Orthopedic Accommodating-feedback Device (ReLOAD) system.
  Interventions: Device: Rehabilitative Lower-limb Orthopedic Accommodating-feedback Device (ReLOAD)
- Amputee Group (Active Comparator): The investigators will recruit a total of 130 subjects (65 at WRNMMC and 65 at the Miami VA) with the goal of consenting and enrolling 100 subjects (50 and WRNMMC and 50 at the Miami VA) with lower limb amputation to utilize the ReLOAD system.
  Interventions: Device: Rehabilitative Lower-limb Orthopedic Accommodating-feedback Device (ReLOAD)

INTERVENTIONS:
Device: Rehabilitative Lower-limb Orthopedic Accommodating-feedback Device (ReLOAD) — The study will use a novel piece of technology, the ReLOAD, which is a data collector system that uses instrumented insoles, custom, miniature (1"x1") microcontroller with accelerometer, gyroscopes, and geomagnetic sensors connected to a Bluetooth transceiver to collect and transmit gait kinematic data to mobile devices, such as an iPad and iPod. When a person walks or performs a specific activity, the ReLOAD system captures the movement, which can then be stored locally within the mobile device and/or encrypted and sent to a secured central server. This allows the patient or provider to access clinically relevant biomechanical data to help guide rehabilitation.

SUMMARY:
This joint research project between the Department of Veterans Affairs (VA) and Department of Defense (DoD) will demonstrate that the implementation of the Mobile Device Outcomes-based Rehabilitation Program (MDORP) will improve the quality of rehabilitative care at a decreased cost to the healthcare system and a reduced burden for service members (SMs) and veterans with lower limb loss. The development of the MDORP will be executed by a multisite translational clinical care team that will use web-based mobile computing devices designed to assess mobility, enable remote prescription of targeted exercise program, and provide continual measureable outcomes to document the continuum of care with the intent of maximizing prosthetic performance while minimizing adverse medical events. The information obtained from this web-based mobile device application will be used by clinicians to promote continuity of care from the DoD and VA facilities nationwide to the community and at home.

ELIGIBILITY:
The following inclusion and exclusion criteria will be used to determine eligibility for the veterans with lower limb loss to participate in the study at the Miami VA and SMs at WRNMMC.

Inclusion Criteria:

* DEERS eligible Veterans/SMs with major unilateral or bilateral lower limb loss at the Symes, Transtibial, Knee Disarticulation, and/or Transfemoral amputation levels
* At least 3 months from initial prosthetic fitting and cleared for at home prosthetic use.
* Male and Females between 20 - 80 years of age
* Determined to be medically stable before participation in the study
* Currently have a well-fitting and properly aligned prosthesis
* Can independently perform exercises at home
* Demonstrate basic proficiency with use of tablet technology

Exclusion criteria:

* Spinal cord injury or lower limb paralysis
* Complete or partial peripheral nerve injury limiting physical performance or increase risk of injury
* Cognitively unable to complete the self-report questionnaires or use tablet technology
* No valid contact information
* Amputation of only toes or upper limb only
* Amputation of upper and lower limb
* The subject is deemed as living too far away for the physical therapist to conduct home visits.
* Evidence of any nerve or brain disorders that affect motion
* Unable to speak or understand English
* The subject does not have the capacity to provide consent.

The following inclusion and exclusion criteria will be used to determine eligibility for the CONTROL subjects to participate in phase I of the study at WRNMMC.

Inclusion Criteria:

* DEERS Eligible males and females between 20-65 years of age
* Determined to be medically stable before participation in the study
* No history of upper or lower limb loss

Exclusion Criteria:

* Evidence of paralysis or other lower limb dysfunction.
* Complete or partial peripheral nerve injury limiting physical performance or increase risk of injury
* Cognitively unable to follow study instructions
* Amputation of upper or lower limb
* Unable to walk 100 meters without an assistive device (cane, walker, etc)
* History of cardiovascular disease that would limit ambulation 100 meters
* Reported symptoms of chest pain or shortness of breath
* Evidence of any nerve or brain disorders that affect motion
* Unable to speak or understand English
* The subject does not have the capacity to provide consent.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-05; Primary Completion 2019-06 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Change in Timed Up and Go (TUG) | Baseline; Weeks 2,4,6 and 8; Month 3 Follow-Up
  The TUG is a measure of basic mobility that assesses the time to complete a sit to stand activity from a standard height chair, ambulate less than 10 feet, perform a turning activity, ambulate back to the chair and perform stand to sit activity. It is a measure of mobility and predictor of falls risk.
Change in Six-minute Walk Test (6MWT) | Baseline; Weeks 2,4,6 and 8; Month 3 Follow-Up
  The 6MWT has been found to be a measure of overall mobility and physical functioning in the lower limb amputee population and geriatric population. It will be used to provide an overall measure of mobility and musculoskeletal endurance.
Change in Amputee Mobility Predictor (AMP) | Baseline; Weeks 2,4,6 and 8; Month 3 Follow-Up
  The AMP is a 21 item clinical tool that assesses current functional capability and mobility with a prosthesis when performing basic daily activities. The AMP assesses the ability of an amputee to complete 20 different items that progress in level of difficulty. Higher AMP scores indicate greater prosthetic ambulation capabilities.
Change in Bilateral-Amputee Mobility Predictor (BAMP) | Baseline; Weeks 2,4,6 and 8; Month 3 Follow-Up
  The BAMP is the AMP adapted for those with bilateral lower limb loss.
Change in Comprehensive High-level Activity Mobility Predictor (CHAMP) | Baseline; Weeks 2,4,6 and 8; Month 3 Follow-Up
  The CHAMP is a clinical tool that assesses an individual's capabilities in performing high-level mobility and agility activities in multiple planes of motion. It consists of four tests (Single Limb Stance, Edgren Side Step Test, T-Test, and Illinois Agility Test) and generates a total score that indicates greater high-level mobility capabilities.
Change in Symmetry of External Work (SEW) | Baseline; Weeks 2,4,6 and 8; Month 3 Follow-Up
  The SEW is a biomechanical outcome measure for assessing dynamic movement symmetry during functional activities. SEW values represent the effort undertaken by each lower-limb in moving the body forward during walking. It will be assessed simultaneously with the TUG, AMP, 6MWT, and CHAMP.
Change in Modified Test of Sensory Integration and Balance (mCTSIB) | Baseline; Weeks 2,4,6 and 8; Month 3 Follow-Up
  The mCTSIB is a test to describe postural control under various sensory conditions. The test requires subjects to maintain balance for 30 seconds in four conditions: firm surface with eyes open, firm surface with eyes closed, standing on foam with eyes open, and standing on foam with eyes closed.

SECONDARY OUTCOMES:
Charleson Co-Morbidity Index | Baseline; Weeks 2,4,6 and 8; Month 3 Follow-Up
  Description of Current Medical Conditions
Bandura's Self-efficacy Survey | Baseline; Weeks 2,4,6 and 8; Month 3 Follow-Up
  Self-motivation for exercise
New Injury Severity Score | Baseline; Weeks 2,4,6 and 8; Month 3 Follow-Up
  History of the musculoskeletal injuries due to the participant's traumatic event will be documented using self-report and past and current medical records from each participant. The injuries will be categorized into anatomical body regions using the Abbreviated Injury Scale (AIS). The New Injury Severity Score (NISS) will be calculated using the AIS for each participant to determine injury severity.
Patient Reported Outcome Measure Information System (PROMIS) | Baseline; Weeks 2,4,6 and 8; Month 3 Follow-Up
  Physical Function domains will be used to describe the participant's performance of standard activities of daily living, pain intensity, pain severity, fatigue with activities, and sleep disturbance. The PROMIS Mental Health domains will be used to describe the participant's current state of depression, anger, and anxiety with daily activities.
International Physical Activity Questionnaire (IPAQ) | Baseline; Weeks 2,4,6 and 8; Month 3 Follow-Up
  Physical Activity Questionnaire
Trinity Amputation and Prosthesis Experience Scale-Revised (TAPES-R) | Baseline; Weeks 2,4,6 and 8; Month 3 Follow-Up
  The TAPES will be administered to the participants with lower limb loss in order to assess psychosocial adjustment, activity restriction, and satisfaction with their current prosthesis. It contains 33 self-reported items; psychosocial adjustment, 15 items; activity restriction, 10 items; and satisfaction, 8 items.
Prosthetic Limb Users Survey- Mobility (PLUS-M) | Baseline; Weeks 2,4,6 and 8; Month 3 Follow-Up
  The PLUS-M is a self-report measure of mobility designed for prosthetic limb users to assess mobility performing different activities of daily living within the home and community.
Socket Fit Comfort Scale | Baseline; Weeks 2,4,6 and 8; Month 3 Follow-Up
  Socket comfort and fit assessment.
Activities-specific balance confidence scale (ABC) | Baseline; Weeks 2,4,6 and 8; Month 3 Follow-Up
  Measurement of balance confidence.
Modified Oswestry Low Back Pain Disability Index (MODI) | Baseline; Weeks 2,4,6 and 8; Month 3 Follow-Up
  The MODI is a 10-item questionnaire that will be used to assess current presence and severity of low back pain with different daily activities.
Lower Extremity Functional Scale (LEFS) | Baseline; Weeks 2,4,6 and 8; Month 3 Follow-Up
  The LEFS is a 20- item questionnaire that assesses one's ability to perform activities of daily life, functional mobility, balance, coordination, and range of motion/strength. It is scored on a 4 point scale for each question for a maximum score of 80.
Height | Baseline
  Height in inches of participant will be collected.
Weight | Baseline
  Weight in kilograms of the participant will be collected.
Body Mass Index | Baseline
  Body Mass Index will be calculated for each participant using their height and weight.
Waist Circumference | Baseline
  Waist Circumference in centimeters will be collected from each participant.
Hip Circumference | Baseline
  Hip Circumference in centimeters will be collected from each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Paul F Pasquina, MD, Principal Investigator — Walter Reed National Military Medical Center, Uniformed Services Univesrity of the Health Sciences, Center for Rehabilitation Sciences Research
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gaunaurd I, Kristal A, Horn A, Krueger C, Muro O, Rosenberg A, Gruben K, Kirk-Sanchez N, Pasquina P, Gailey R. The Utility of the 2-Minute Walk Test as a Measure of Mobility in People With Lower Limb Amputation. Arch Phys Med Rehabil. 2020 Jul;101(7):1183-1189. doi: 10.1016/j.apmr.2020.03.007. Epub 2020 Apr 6. PMID 32272105